CLINICAL TRIAL: NCT02228174
Title: Evaluation of the Gynesonics System for Transcervical Treatment of Symptomatic Uterine Fibroids With Radiofrequency Ablation Under Integrated Intrauterine Sonography Guidance
Brief Title: Sonography Guided Transcervical Ablation of Uterine Fibroids
Acronym: SONATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynesonics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL04502
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Menorrhagia
Keywords: Abnormal Uterine Bleeding associated with fibroids; AUB-L; Fibroids; Heavy menstrual bleeding; HMB; Myoma; Menorrhagia
MeSH Terms: conditions — Menorrhagia; Leiomyoma; Myoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Subjects Treated with Sonata (Experimental): Intervention: Intrauterine Ultrasound-Guided Radiofreq. Ablation System or the Sonata, which is a sonography guided transcervical ablation device intended for treatment of symptomatic uterine fibroids. Subjects with symptomatic uterine fibroids and heavy menstrual bleeding who met the study population selection criteria received treatment with Sonata.
  Interventions: Device: Intrauterine Ultrasound-Guided Radiofreq. Ablation System

INTERVENTIONS:
Device: Intrauterine Ultrasound-Guided Radiofreq. Ablation System — The Sonata System combines intrauterine ultrasound (IUUS) with radiofrequency (RF) ablation in a single handpiece. Sonata is suitable in an inpatient or outpatient setting, and is intended for diagnostic intrauterine imaging and transcervical treatment of symptomatic uterine fibroids, including those associated with heavy menstrual bleeding(HMB).
  Other Names: Gynesonics Sonata System

SUMMARY:
The objective of this study is to establish the safety and effectiveness of the Sonata® System in the treatment of symptomatic uterine fibroids.

DETAILED DESCRIPTION:
In this single-arm study, subjects who have symptomatic uterine fibroids will have transcervical RF ablation of uterine fibroids under intrauterine ultrasound guidance using the Gynesonics Sonata System.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal
* ≥ 25 and ≤ 50 years of age at time of enrollment
* experienced heavy menstrual bleeding associated with fibroids (AUB-L) for at least 3 months
* between 1-10 fibroids of FIGO types 1, 2, 3, 4, and/or type 2-5, with diameter ≥ 1.0 cm and ≤ 5.0 cm
* at least one type 1, type 2, type 3, or type 2-5 fibroid.
* PBAC score ≥ 150 and ≤ 500
* consistent menstrual cycles
* not at material risk for pregnancy
* speaks and reads a language for which validated questionnaires are available
* willing and able to read, understand, and sign the informed consent form, to participate in the study and to adhere to all study follow-up requirements

Exclusion Criteria:

* pregnancy
* urgent need for surgery to treat fibroid symptoms
* desire for current or future childbearing
* presence of a tubal implant for sterilization
* postmenopausal by history
* presence of type 0 fibroids, unless < 1 cm in diameter
* presence of a single polyp ≥ 1.5 cm, or multiple polyps of any size
* any fibroid of FIGO type 1, type 2, type 3, type 4, or type 2-5 with diameter > 5.0 cm
* bulk symptoms in the presence of one or more fibroids of FIGO type 5, type 6, or type 7
* exclusive presence of fibroids that are insufficient to explain the severity of symptoms
* presence of clinically relevant fibroids that cannot be treated for technical reasons
* presence of an extrauterine pelvic mass that has not been diagnosed as benign
* IUD/IUS in situ within the washout period
* previous procedure for fibroids or heavy menstrual bleeding other than myomectomy
* myomectomy within 12 months
* any abnormality of the endometrial cavity that obstructs access of the handpiece
* contraindication to MRI
* total uterine volume > 1000 cc
* clinically significant adenomyosis
* confirmed or suspected diagnosis of clinically relevant endometriosis
* one or more clinically relevant fibroids that are significantly calcified.
* previous pelvic irradiation
* renal insufficiency [serum creatinine ≥ 1.5 mg/dL (132.6 μmol/L)]
* evidence of disorders of hemostasis (AUB-C)
* abnormal cervical cytology that is unevaluated or untreated in adherence with national guidelines
* endometrial hyperplasia (AUB-M), including simple hyperplasia without atypia
* confirmed abdominal / pelvic malignancy within the previous five years
* active pelvic infection or current positive testing for pelvic gonorrhea or chlamydia;
* use of a hormonally-relevant medication within the washout period
* use of an antifibrinolytic agent while undergoing any screening procedures
* current use of anticoagulant therapy
* chronic pelvic pain (disruptive for at least six months) or significant baseline pelvic or menstrual pain
* chronic uncontrolled moderate and severe hypertension
* hypoplastic or otherwise short uterus
* major medical or psychiatric illness or other factors that may affect general health or subject's ability to adhere to the follow-up schedule or provide valid subject self-assessment data
* any other reason for which the individual study subject is not appropriate or suitable for participation

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2014-10; Primary Completion 2017-10-18 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (22):
  - Kelly H. Roy M.D. P.C., Phoenix, Arizona
  - Advanced Women's Health Institute, Denver, Colorado
  - Christiana Care Health Services, Inc., Newark, Delaware
  - George Washington University Hospital, Washington D.C., District of Columbia
  - KO Clinical Research, LLC, Fort Lauderdale, Florida
  - Visions Clinical Research, Wellington, Florida
  - The Advanced Gynecologic Surgery Institute - Charles E. Miller, MD & Associates, Naperville, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Wayne State University, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Clinic, Minimally Invasive Gynecology, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Basque Women's Care, Albuquerque, New Mexico
  - Montefiore Medical Center, New York, New York
  - Carolina Women's Research and Wellness Center, Durham, North Carolina
  - Drexel University, Philadelphia, Pennsylvania
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - Baylor Research Institute, Fort Worth, Texas
  - Willowbend Health and Wellness Associates, Frisco, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Hospital Universitario "Dr. José Eleuterio González" de la Universidad Autónoma de Nuevo León, Monterrey, N.L., Mexico

REFERENCES:
- [Derived] Christoffel L, Bends R, Toub D, Schiermeier S, Pschadka G, Engelhardt M, Quinn S, Hartmann M, Habiba M, Felberbaum R, Brossner A, Schippert C, Romer T. Pregnancy Outcomes After Transcervical Radiofrequency Ablation of Uterine Fibroids with the Sonata System. J Gynecol Surg. 2022 Jun 1;38(3):207-213. doi: 10.1089/gyn.2021.0136. Epub 2022 Jun 13. PMID 35785107
- [Derived] Roy K, Robinson JK. Durable Improvement in Generic and Fibroid-Specific Quality of Life in Women Treated with Transcervical Fibroid Ablation with the Sonata System After Three Years. J Gynecol Surg. 2022 Apr 1;38(2):143-147. doi: 10.1089/gyn.2021.0073. Epub 2022 Apr 1. PMID 35497488
- [Derived] Shifrin G, Engelhardt M, Gee P, Pschadka G. Transcervical fibroid ablation with the Sonata system for treatment of submucous and large uterine fibroids. Int J Gynaecol Obstet. 2021 Oct;155(1):79-85. doi: 10.1002/ijgo.13638. Epub 2021 Mar 17. PMID 33544889
- [Derived] Chudnoff S, Guido R, Roy K, Levine D, Mihalov L, Garza-Leal JG. Ultrasound-Guided Transcervical Ablation of Uterine Leiomyomas. Obstet Gynecol. 2019 Jan;133(1):13-22. doi: 10.1097/AOG.0000000000003032. PMID 30531573

RESULTS

PARTICIPANT FLOW:
Groups:
- Sonata: Subjects treated with the Sonata System.
Period: Overall Study
Arm/Group | Sonata
Started | 147
Full Analysis Population | 143 (Subjects who didn't become pregnant or diagnosed with an interfering medical condition at 12-months)
Completed | 142
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population was comprised of subjects who were treated and had any post-baseline data.
Groups:
- Sonata: Subjects treated with Sonata System.
Arm/Group | Sonata
Number analyzed (Participants) | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (4.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 43
  Black or African American | 49
  White | 60
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 125
  Mexico | 22
Pictorial Blood Loss Assessment Chart [Mean (Standard Deviation); unit: Index] — The PBAC is a validated assessment tool to estimate menstrual blood loss using icons representing various degrees of saturation of sanitary products. It is not a scale, but rather an index with values ≤100 to have been reported to represent eumenorrhea. In this study, women had to have heavy menstrual bleeding marked by a baseline PBAC of >=150 and <=500 to be eligible for study participation.
  Index | 300.6 (98.47)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With ≥ 50% Reduction in Menstrual Blood Loss as Assessed by Pictorial Blood Loss Assessment Chart (PBAC)
Description: The proportion of subjects with a minimum of 50% reduction in menstrual blood loss at 12 months post-procedure compared to baseline as assessed by PBAC. Success for individual subjects was defined as a ≥ 50% reduction from baseline in menstrual blood loss and a final PBAC score < 250. Endpoint success was defined as the lower confidence limit of the percentage of subject success ≥ 45%. The PBAC is a validated tool used to diagnose heavy menstrual bleeding and track menstrual bleeding. Women were asked to record daily use of tampons and sanitary towels by placing a tally mark under the day next to the box that represented how stained the sanitary materials were each time they were changed during the menstrual cycle. The tally marks were added up depending on the saturation level to provide a score. The score does not have an upper limit as it is not a "scale". PBAC ≥ 150 is associated with heavy menstrual bleeding.
Time Frame: Baseline and 12 Months
Population: Full Analysis Population (143) minus 1 subject who had surgical reintervention prior to 12 months and was excluded from analysis of bleeding reduction coprimary endpoint per the Statistical Analysis Plan.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Subjects Treated With Sonata: Sonata is a sonography guided transcervical ablation device intended for treatment of symptomatic uterine fibroids. Subjects with symptomatic uterine fibroids and heavy menstrual bleeding who met the study population selection criteria received treatment with the Sonata system.
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 142
percentage of participants | 64.8 [56.3 to 72.6]

2. Primary Outcome: Percentage of Subjects Without Surgical Re-intervention for Heavy Menstrual Bleeding Due to Treatment Failure
Description: This endpoint computed the rate of not having a surgical reintervention for heavy menstrual bleeding due to treatment failure. As the success criterion for this endpoint was "no surgical reintervention for HMB due to treatment failure at 12 months", the endpoint assessed the rate of subjects without surgical reintervention success due to treatment failure within the 12-month post-treatment period. Rate was calculated using the life-table method.
Time Frame: 12 Months
Population: Full Analysis Population (143 subjects)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 143
Percentage of Participants | 99.3 [95.1 to 99.9]

3. Secondary Outcome: Safety - Percentage of Subjects With Adverse Device Effects (Serious or Non-serious)
Description: Procedure safety was assessed by recording all adverse device effects that occured during or subsequent to treatment on the day of the procedure. Longer-term safety was assessed by recording any untoward medical occurrence since baseline at each follow-up visit.
Time Frame: Each Follow-up Visit through 24 Months
Population: Safety population - all subjects who recieved the Sonata treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 147
Participants | 0

4. Secondary Outcome: Percentage Change in Total and Perfused Mean Maximal Fibroid Volumes at 12 Months
Description: The percent change in total and perfused volume of dominant fibroid were determined by comparing contrast-enhanced MRI at baseline and at 12 months.
Time Frame: Baseline and 12 Months
Population: Full Analysis Population without imputation for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 129
percentage change
  % Change in Total Mean Maximal Fibroid Volume | -62.4 (32.81)
  % Change in Perfused Mean Maximal Fibroid Volume: number analyzed (Participants) | 128
  % Change in Perfused Mean Maximal Fibroid Volume | -63.9 (31.44)

5. Secondary Outcome: Change in the Symptom Severity Score (SSS) and Quality of Life (HR-QoL) Subscales of the Uterine Fibroid Symptom and Quality of Life (UFS-QoL) Questionnaire at 12 Months
Description: The Symptom Severity Score (SSS) and Health-Related Quality of Life Score (HR-QoL) are calculated from a subset of the Uterine Fibroid Symptom and Quality of Life (UFS-QoL) questionnaire, a validated and fibroid-specific assessment tool. The UFS-QoL is a uterine fibroid-specific questionnaire developed to evaluate the symptoms of uterine fibroids and their impact on quality of life related to health. SSS and HR-QoL subscale scores are summed and transformed into a 0-100 point scale. The SSS and HR-QoL subscale scores are inversely related with higher SSS indicating greater symptoms while higher HR-QoL scores indicate better quality of life.
Time Frame: Baseline and 12 Months
Population: Full Analysis Population without imputation for this outcome measure.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 135
points on a scale
  Mean Change in SSS at 12 Months | -32.1 (21.03)
  Mean Change in HR-QoL at 12 Months: number analyzed (Participants) | 134
  Mean Change in HR-QoL at 12 Months | 43.7 (24.25)

6. Secondary Outcome: Time to Return to Normal Activity (RTNA) in Days
Description: Subjects were given a questionnaire at discharge and asked to daily respond to the questionnaire on whether or not they returned to normal activities.
Time Frame: 30 Day post-procedure
Population: Full Analysis Population without imputation for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 139
Days | 2.2 (2.23)

7. Secondary Outcome: Overall Treatment Effect (OTE) at 12 Months
Description: The Overall Treatment Effect is a questionnaire for subjects to report their perceived treatment benefit at a given timepoint as either improved, no change, or worsened.
Time Frame: 12 Months
Population: Full Analysis Population without imputation for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 135
Participants
  Fibroid Symptoms Improved | 130
  Fibroid Symptoms Unchanged | 4
  Fibroid Symptoms Worsened | 1

8. Secondary Outcome: Subject Satisfaction With Treatment at 12 Months
Description: Subjects were asked to rate their level of satisfaction with the treatment. The possible ratings were as follows: "very satisfied", "moderately satisfied", "somewhat satisfied", "somewhat dissatisfied", "moderately dissatisfied", and "very dissatisfied".
Time Frame: 12 Months
Population: Full Analysis Population without imputation for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 135
Participants
  Very Satisfied | 95
  Modeately Satisfied | 24
  Somewhat Satisfied | 12
  Somewhat Dissatisfied | 3
  Moderately Dissatisfied | 1
  Very Dissatisfied | 0

9. Secondary Outcome: Subject Willingness to Recommend Procedure at 12 Months
Description: Subjects were asked whether they would recommend the procedure to a friend with the same health problems. The possible responses were: "definitely yes", "probably yes", "probably no", and "definitely no".
Time Frame: 12 Months
Population: Full Analysis Population without imputation for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 135
Participants
  Definitely Yes | 110
  Probably Yes | 21
  Probably No | 4
  Definitely No | 0

10. Secondary Outcome: Change in General Health State at 12 Months
Description: Change in general health state was assessed with the EuroQOL EQ-5D. The EQ-5D is a standardized instrument for use as a measure of health outcome. Applicable to a wide range of health conditions and treatments, EuroQOL EQ-5D provides a simple descriptive profile and a single index value for health status. The EQ-5D consists of five questions that provide a description of the patient's health state with scores ranging from 0 (indicating death) to 1 (indicating perfect health). An increase of 0.04 in EQ-5D is considered by health economists to represent a minimally important difference.
Time Frame: Baseline and 12 Months
Population: Full Analysis Population without imputation for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 133
units on a scale | 0.17 (0.223)

11. Secondary Outcome: Subject Pain
Description: Prior to discharge, subjects were asked to rate their experience of pain using a pain Visual Analog Scale (VAS). The VAS for pain is a measurement instrument by which subjects report the intensity of their pain with a quantitative value from 0 (no pain) to 10 (worst pain ever).
Time Frame: Immediately Post-procedure as well as Pre-discharge (Day 0)
Population: Safety Population - all treated subjects (147).
Measure: Mean (Standard Deviation); unit: score on a scale from 0 to 10
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 147
score on a scale from 0 to 10
  Overall Pain During Procedure | 0.24 (0.948)
  Overall Pain During Recovery | 2.63 (2.771)

12. Secondary Outcome: Procedure Tolerance
Description: Prior to discharge, subjects were asked to rate their tolerance of the procedure. The possible responses were "very tolerable", "moderately tolerable", "minimally tolerable", "intolerable".
Time Frame: Post-procedure (Day 0)
Population: Safety Population - all treated subjects (147).
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 147
Participants
  Very Tolerable | 95
  Moderately Tolerable | 45
  Minimally Tolerable | 4
  Intolerable | 3

13. Secondary Outcome: Mean Length of Stay
Description: Length of stay (in hours) was assessed by recording the duration from the start of the procedure to discharge.
Time Frame: Day 0 - Day of Treatment
Population: Safety Population - all treated subjects (147).
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 147
Hours | 2.54 (1.243)

14. Secondary Outcome: Occurrence of Pregnancy
Description: Subjects were asked about the possible occurrence of pregnancy.
Time Frame: All Follow-up Visits through 24 Months
Population: Full Analysis Population (143 subjects).
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 143
Participants | 1

15. Secondary Outcome: Pregnancy Outcome - Gestation Age
Description: If pregnancy occurred during the study follow-up period, information regarding gestation age was collected.
Time Frame: 24 Months
Population: 1 subject with pregnancy
Measure: Number; unit: weeks
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 1
weeks | 38.2

16. Secondary Outcome: Pregnancy Outcome - Birth Weight
Description: If pregnancy occurred during the study follow-up period, information regarding birth weight was collected.
Time Frame: 24 Months
Population: 1 subject with pregnancy
Measure: Number; unit: grams
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 1
grams | 4005

17. Secondary Outcome: Change in Work Productivity and Activity Impairment Due to Uterine Fibroid Symptoms at 12 Months
Description: The Work Productivity and Activity Impairment questionnaire for a specific health problem (WPAI:SHP) is a standardized instrument for making a quantitative assessment of work impairment and activity impairment attributable to a specific health problem (WPAI:SHP). The assessments are expressed in percentages. The endpoint assessed the difference in these percentages from baseline to 12 months.
Time Frame: Baseline and 12 Months
Population: Subset of the Full Analysis Population who were employed and had paired responses at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Subjects Treated With Sonata
Number analyzed (Participants) | 112
percentage change
  Change in mean Overall Work Impairment: number analyzed (Participants) | 81
  Change in mean Overall Work Impairment | -40.0 (34.22)
  Change in mean Activity Impairment: number analyzed (Participants) | 105
  Change in mean Activity Impairment | -46.2 (31.21)

ADVERSE EVENTS:
Time Frame: 12 Months
Description: All Adverse Events were evaluated by the Sponsor and reviewed by the study's Medical Advisory Board for relatedness and seriousness.
Arm/Group | Sonata
All-Cause Mortality (participants affected / at risk) | 0/147
Serious Adverse Events (participants affected / at risk) | 2/147
Other Adverse Events (participants affected / at risk) | 60/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sonata (N=147)
Deep Vein Thrombus (Vascular disorders) | 1 (1)
Vaginal Discharge with Overnight Hospital Stay (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sonata (N=147)
Cramping/Pain (Reproductive system and breast disorders) | 11 (12)
Fibroid Shedding (Reproductive system and breast disorders) | 45 (53)
Genitourinary Infections (Infections and infestations) | 7 (8)
Vaginal Discharge (Reproductive system and breast disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT02228174/Prot_000.pdf
  • Statistical Analysis Plan (2014-09-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT02228174/SAP_001.pdf